CLINICAL TRIAL: NCT04386278
Title: RI.2 OrthoPulse Gen 2 Initial Device Evaluation and Assessment of Clinical
Brief Title: OrthoPulse Gen 2 Initial Device Evaluation and Assessment of Clinical Effectiveness (CA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped because slow enrolment.
Sponsor: Biolux Research Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RI.2
Record Dates: First submitted 2020-04-08; First posted 2020-05-13 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Orthodontic Tooth Movement

STUDY DESIGN:
Intervention Model Description: Each group in this study includes a different device iteration that is being investigated in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Intervention 1 (Experimental): Side one: No treatment Side two: OrthoPulse Gen 2 (2RP) for one minute
  Interventions: Device: Intervention 1
- Intervention 2 (Experimental): Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (2RP) for one minute
  Interventions: Device: Intervention 2
- Intervention 3 (Experimental): Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (2RP) for 5 minutes
  Interventions: Device: Intervention 3
- Intervention 4 (Experimental): Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (2RCW) for five minutes
  Interventions: Device: Intervention 4
- Intervention 5 (Experimental): Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (3RB 2RL) for one minute
  Interventions: Device: Intervention 5
- Intervention 6 (Experimental): Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (3RB 2RL) for five minutes
  Interventions: Device: Intervention 6
- Intervention 7 (Experimental): Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (3RB 2RL) for one minute
  Interventions: Device: Intervention 7
- Intervention 8 (Experimental): Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (3RB 2RL) for five minutes
  Interventions: Device: Intervention 8

INTERVENTIONS:
Device: Intervention 1 — Side one: No treatment Side two: OrthoPulse Gen 2 (2RP) for one minute
  Arms: Intervention 1
Device: Intervention 2 — Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (2RP) for one minute
  Arms: Intervention 2
Device: Intervention 3 — Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (2RP) for 5 minutes
  Arms: Intervention 3
Device: Intervention 4 — Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (2RCW) for five minutes
  Arms: Intervention 4
Device: Intervention 5 — Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (3RB 2RL) for one minute
  Arms: Intervention 5
Device: Intervention 6 — Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (3RB 2RL) for five minutes
  Arms: Intervention 6
Device: Intervention 7 — Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (3RB 2RL) for one minute
  Arms: Intervention 7
Device: Intervention 8 — Side one: OrthoPulse (approved device) Side two: OrthoPulse Gen 2 (3RBP) for five minutes
  Arms: Intervention 8

SUMMARY:
This is a prospective, interventional, non-randomized, control, split-mouth, open-label, single centre, private practice study aimed to evaluate the effect of tooth movement during orthodontic treatment using a removeable thermoplastic orthodontic appliance. Intrusion and extrusion will be conducted using bilaterally equivalent elastomeric forces of 50 grams.

A comparison of the rate of bilateral orthodontic tooth movement will be conducted using six (6) varied photobiomodulation interventions on the maxillary (upper) and mandibular (lower) arches. The OrthoPulse Gen 2 and OrthoPulse (commercially approved) devices are being used in this clinical investigation. Each subject enrolled will go through intrusion and extrusion.

All subjects will be allocated to an OrthoPulse split-mouth intervention by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 19 years of age or older
* Likely to be compliant to OrthoPulse use, aligner wear, and Dental Monitoring scanning
* Have a compatible iOS or Android device and are willing to download the OrthoPulse and Dental Monitoring apps for frequent automatic syncing of data

Exclusion Criteria:

* Patient is currently enrolled in another clinical study
* Crowding or rotations of bilateral bicuspids that would prevent or interfere with intrusion
* Periodontally involved teeth, acute oral infection or periodontal disease
* Patient has active/untreated caries
* Use of bisphosphonates at any time
* Use of drugs that may cause photosensitivity
* History of photosensitivity
* Epilepsy
* Pregnant or planning pregnancy during the study.
* Patient plans to relocate over the treatment period

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
The rate of orthodontic tooth movement | 36 days (±12 days) from T0 visit
  The rate of orthodontic tooth movement during intrusion at 36 days (±12 days) from the T0 Visit (measured in mm per week).

SECONDARY OUTCOMES:
Peak Pain: Questionnaire | 7 Days
  Assess peak pain experienced over first seven (7) days of treatment during intrusion using a questions similar in nature to a Visual Analog Scale (subject to complete pain questionnaire).
Root Resorption | 36 days (±12 days) from T0 visit
  Assess tooth resorption by measuring the root length of the first or second bicuspid bilaterally from baseline to T3
Initial Safety of Device | From enrolment to study completion, anticipated six (6) months
  Confirmation of safety through collection of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Peter Brawn, Vancouver, B.C, Canada

IPD SHARING:
Plan to Share IPD: No